CLINICAL TRIAL: NCT00917293
Title: A Randomized, Double-Blind, Placebo-Controlled, Comparative Study to Evaluate the Safety and Efficacy of Pyridoxal 5' -Phosphate in the Treatment of Tardive Dyskinesia in Patients With Schizophrenia and Schizoaffective Disorders
Brief Title: Safety and Efficacy of Pyridoxal 5' -Phosphate in the Treatment of Tardive Dyskinesia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: modified formulation under investigation
Sponsor: Medicure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08030
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Tardive Dyskinesia
Keywords: Tardive Dyskinesia; Schizophrenia; Pyridoxal 5'-phosphate
MeSH Terms: conditions — Tardive Dyskinesia; Schizophrenia | interventions — Pyridoxal Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pyridoxal 5'-Phosphate (Experimental): Pyridoxal 5'-Phosphate, enteric-coated 2x 250mgs po bid.
  Interventions: Drug: Pyridoxal 5'-Phosphate
- Placebo (Placebo Comparator): Placebo 2 pills, po bid.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyridoxal 5'-Phosphate — Pyridoxal 5'-Phosphate 500mgs po bid for 12 weeks.
  Other Names: Tardoxal
  Arms: Pyridoxal 5'-Phosphate
Drug: Placebo — Placebo 2 pills, po bid.
  Arms: Placebo

SUMMARY:
The primary objective is to assess the safety and effectiveness of Pyridoxal 5'-Phosphate on the reduction of expressed symptoms of tardive dyskinesia in patients with schizophrenia and schizoaffective disorders.

DETAILED DESCRIPTION:
This study will assess the effect of Pyridoxal 5'-Phosphate on the reduction of expressed symptoms of moderate to severe tardive dyskinesia in patients with schizophrenia and schizoaffective disorders who are on a stable dose, and regime, of either a long acting (i.e. depot/IM) or oral antipsychotic medication, as compared to placebo.

Symptoms will be assessed through the administration and scoring of Abnormal Involuntary Movement Scale (AIMS), specifically on items 1 through 7 (facial and oral movements, extremity movements and trunk movements) at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed an informed consent document indicating that they understand the purpose of the study, its objectives, and the expectations of participation in the study and that they agree to participate in the study.
2. Meet current diagnostic criteria for Schizophrenia (Disorganized [295. 10], Paranoid [295.30], or Residual [295.60]), or Schizoaffective Disorder [295.70] as defined by the DSM-IV for at least 3 months before screening.
3. Have been on a stable dose and regime of a LAI for at least 3 injection intervals or oral antipsychotic for at least 1 month prior to randomization and are expected to remain on this stable dose and regime throughout their participation in the study.
4. Meet current diagnostic criteria for Neuroleptic Induced Tardive Dyskinesia [333.82] as defined by the DSM-IV.
5. Scoring ≥3 (moderate) on item 8, the "severity of abnormal movements overall" section of the AIMS.
6. Score ≥3 (moderate) on at least one item, or ≥2 (mild) on at least 2 items, and an overall total score of ≥5 on items 1 through 7 (facial and oral movements, extremity movements and trunk movements) sections of the AIMS.
7. Female patients must be post-menopausal for at least 2 years or surgically sterile. Women of childbearing potential must be using or agree to use a reliable form of contraception before entry into and during participation in the study. Reliable contraception can include an oral or other hormonal contraceptive started at least 4 weeks prior to randomization, a barrier method such as condoms or a diaphragm used with spermicide, or an intrauterine device (IUD).
8. Patients must be capable of administering study medication themselves or will have assistance with the administration of the study medication consistently available throughout the study.

Exclusion Criteria:

1. Involuntarily committed to a psychiatric hospital or correctional facility.
2. A primary active DSM-IV diagnosis or co-morbid Axis 1 diagnosis other than schizophrenia or schizoaffective disorder.
3. PANSS Score > than 120 at the screening visit.
4. Current medical diagnosis that which could confound the interpretation or evaluation of the indication under study (i.e. Parkinson's Disease, Huntington's Chorea, Muscular Dystrophy, Tourette's Syndrome).
5. History of liver cirrhosis, chronic active hepatitis (known positive serum test within 6 months of enrollment) or severe liver dysfunction, or liver transaminase ≥3 times ULN at screening (or obtained within 30 days prior to screening visit)
6. History of malignancy during the last 5 years.
7. Pregnant or any woman of childbearing potential who is not using a reliable form of contraception (this can include an oral or other hormonal contraceptive started at least 4 weeks prior to randomization, a barrier method such as condoms or a diaphragm used with spermicide, or an intrauterine device (IUD)). Women who have been post-menopausal for at least two years or who have undergone surgical sterilization are considered to be not of childbearing potential.
8. Any medical, such as unstable cardiovascular, respiratory, neurological, renal, hepatic, immunological or endocrine, or psychiatric condition which in the opinion of the investigator makes the patient an unsuitable candidate for the study.
9. History of any pre-existing gastrointestinal narrowing or inability to swallow the oral study medication whole with the aid of water.
10. Male and female patients with a BMI of ≥20.
11. Significant, ongoing alcohol or drug dependency within 3 months before screening as defined by the DSM-IV (nicotine will not be exclusionary).
12. Significant risk of suicide or violent behavior as clinically assessed by the investigator.
13. Participation in any other investigational drug or device study within 30 days of randomization.
14. Patients who have previously participated in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-05; Primary Completion 2012-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be a reduction in the total AIMS score for items 1 through 7 (facial and oral movements, extremity movements and trunk movements) across treatment groups. . | From baseline through to week 12

SECONDARY OUTCOMES:
An AIMS score reduction (items 1-7) across arms over course of study amongst completers; determine whether the proportion of responders differs between treatment arms; a reduction in the AIMS score, items 1 - 7 total, across treatment arms. | From baseline through to Week 12 and Baseline compared to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Gary J. Remington, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (4):
- Canada (3):
  - Vancouver Island Health Authority, Victoria, British Columbia
  - Centre for Addiction and Mental Health, Toronto, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
- Schizophrenia Research Foundation (SCARF) Mental Health Centre, Chennai, Tamil Nadu, India